CLINICAL TRIAL: NCT02485106
Title: Effect of Gut Decontamination Using Rifaximin in the Patients With Severe Alcoholic Hepatitis
Brief Title: Rifaximin Use in Severe Alcoholic Hepatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Do Seon Song, Clinical assistant professor, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDS-SAH-001
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Rifaximin; Adrenal Cortex Hormones; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin group (Active Comparator): Corticosteroid or Pentoxifylline for 28 days Rifaximin 400mg tid for 28 days
  Interventions: Drug: Rifaximin; Drug: Corticosteroid or pentoxifylline
- Control group (Active Comparator): Corticosteroid or Pentoxifylline for 28 days
  Interventions: Drug: Corticosteroid or pentoxifylline

INTERVENTIONS:
Drug: Rifaximin — 400mg three times per day for 28 days
  Arms: Rifaximin group
Drug: Corticosteroid or pentoxifylline — Corticosteroid 40mg/day or pentoxifylline 400mg three times per day for 28 days

SUMMARY:
This study aimed to investigate the effect of decontamination by rifaximin in severe alcoholic hepatitis patients. Patients who take corticosteroid or pentoxifylline will be randomly allocated to rifaximin group or control group.

ELIGIBILITY:
Inclusion Criteria:

* Heavy alcohol drinking within 3 months (Over 40 g/day)
* Maddrey's discriminant function ≥ 32
* AST/ALT ration ≥ 2
* Bilirubin level ≥ 5mg/dL
* Any one of the following additional criteria : hepatic encephalopathy, enlarged, tender liver, or peripheral leucocytosis
* Age : 19-75
* Jaundice within 3 months

Exclusion Criteria:

* Other causes of chronic liver disease (HBV, HCV, or autoimmune hepatitis)
* Antibiotics or probiotics use within 8 weeks
* Drug induced hepatotoxicity
* Acute viral hepatitis (HAV or HEV)
* Hepatic abscess or cholagitis
* Hepatocellular carcinoma of modified UICC stage II, III or IV
* Malignant tumor other than HCC
* Pregnancy
* Severe chronic extrahepatic disease
* Type I hepatorenal syndrome
* Hepatic encephalopathy grade II or IV
* Severe infection

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6-month

REFERENCES:
- [Derived] Song DS, Yang JM, Jung YK, Yim HJ, Kim HY, Kim CW, Kim SS, Cheong JY, Lee HL, Lee SW, Yoo JJ, Kim SG, Kim YS. Rifaximin treatment in patients with severe alcohol-associated hepatitis: A multicenter, randomized controlled, open-label, pilot trial. Ann Hepatol. 2025 Jan-Jun;30(1):101749. doi: 10.1016/j.aohep.2024.101749. Epub 2024 Dec 9. PMID 39662593